CLINICAL TRIAL: NCT05237635
Title: Defining Decision Thresholds for Judgments on Health Benefits and Harms Using the GRADE Evidence to Decision (EtD) Frameworks: Protocol for a Randomized Methodological Study (GRADE-THRESHOLD)
Brief Title: Defining Decision Thresholds for Judgments on Health Benefits and Harms: Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: GRADETHRESHLD
Record Dates: First submitted 2021-12-08; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Decision Support Techniques; GRADE Approach
Keywords: Evidence to Decision framework; Clinical practice guidelines; Evidence-based medicine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Threshold estimates (Experimental): Descriptive case-scenarios
  Interventions: Other: descriptive case-scenarios
- Alternative threshold estimates (Active Comparator): Descriptive case-scenarios
  Interventions: Other: descriptive case-scenarios

INTERVENTIONS:
Other: descriptive case-scenarios — Each case-scenario will include: (1) a GRADE Summary of Finding (SoF) table providing information about the Population, Intervention, Comparator, Outcome (PICO), the relative and absolute anticipated effects of the intervention, and the certainty in the evidence; (2) a Health Outcome Descriptor describing key attributes of the outcome under consideration including symptoms, time horizon, testing and treatment, and consequences; a measure of the impact on health of the outcome (also known as 'value' of the outcome or 'health utility' in health economics).

SUMMARY:
The objective of this study is an approach to derive and use decision-thresholds for judgments on health benefits and harms using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) Evidence to Decision (EtD) frameworks.

DETAILED DESCRIPTION:
The objective of this study is to derive decision-thresholds (DTs) for Evidence to Decision (EtD) judgments on the magnitude of health benefits and harms. The study hypothesis is that DTs could discriminate between the four categories for EtD judgments. Explicit DTs, providing an indication for which could be the appropriate judgment for a given scenario, might have the potential to support panels of decision-makers in their work, facilitate a common understanding, and promote consistency and transparency in judgments.

Study investigators will conduct a methodological randomized controlled trial to collect the data that allow deriving the decision-thresholds. They will invite clinicians, epidemiologists, decision scientists, health research methodologists, experts in Health Technology Assessment (HTA), members of guideline development groups and the public to participate in the trial. Then, investigators will investigate the validity of decision-threshold by measuring the agreement between judgments that were made in the past by guideline panels and the judgments that the DTs approach would suggest if applied on the same guideline data.

ELIGIBILITY:
Inclusion Criteria:

The target population of the survey will include:

* clinicians
* epidemiologist
* decision scientists
* health research methodologists
* experts in health technology assessment (HTA)
* and members of guideline working groups
* members from the general public

Exclusion Criteria:

• Prior participation in the survey

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1406 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Small effect of an intervention | immediate after completion of study
  Questionnaire: Participants will be asked to indicate which decision threshold for discriminating between EtD judgments of 'Trivial or None' and 'Small' they felt appropriate at the time of participation in the survey.
Moderate effect of an intervention | immediate after completion of study
  Questionnaire:Participants will be asked to indicate which decision threshold for discriminating between EtD judgments of 'Small' and 'Moderate' they felt appropriate at the time of participation in the survey.
Large effect of an intervention | immediate after completion of study
  Questionnaire:Participants will be asked to indicate which decision threshold for discriminating between EtD judgments of 'Moderate' and Large' they felt appropriate at the time of participation in the survey.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Standards for Developing Trustworthy Clinical Practice Guidelines; Graham R, Mancher M, Miller Wolman D, Greenfield S, Steinberg E, editors. Clinical Practice Guidelines We Can Trust. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209539/ PMID 24983061
- [Background] Schunemann HJ. Guidelines 2.0: do no net harm-the future of practice guideline development in asthma and other diseases. Curr Allergy Asthma Rep. 2011 Jun;11(3):261-8. doi: 10.1007/s11882-011-0185-8. PMID 21409613
- [Background] Atkins D, Eccles M, Flottorp S, Guyatt GH, Henry D, Hill S, Liberati A, O'Connell D, Oxman AD, Phillips B, Schunemann H, Edejer TT, Vist GE, Williams JW Jr; GRADE Working Group. Systems for grading the quality of evidence and the strength of recommendations I: critical appraisal of existing approaches The GRADE Working Group. BMC Health Serv Res. 2004 Dec 22;4(1):38. doi: 10.1186/1472-6963-4-38. PMID 15615589
- [Background] Alonso-Coello P, Schunemann HJ, Moberg J, Brignardello-Petersen R, Akl EA, Davoli M, Treweek S, Mustafa RA, Rada G, Rosenbaum S, Morelli A, Guyatt GH, Oxman AD; GRADE Working Group. GRADE Evidence to Decision (EtD) frameworks: a systematic and transparent approach to making well informed healthcare choices. 1: Introduction. BMJ. 2016 Jun 28;353:i2016. doi: 10.1136/bmj.i2016. No abstract available. PMID 27353417
- [Background] Alonso-Coello P, Oxman AD, Moberg J, Brignardello-Petersen R, Akl EA, Davoli M, Treweek S, Mustafa RA, Vandvik PO, Meerpohl J, Guyatt GH, Schunemann HJ; GRADE Working Group. GRADE Evidence to Decision (EtD) frameworks: a systematic and transparent approach to making well informed healthcare choices. 2: Clinical practice guidelines. BMJ. 2016 Jun 30;353:i2089. doi: 10.1136/bmj.i2089. No abstract available. PMID 27365494
- [Background] Marcucci M, Sinclair JC. A generalised model for individualising a treatment recommendation based on group-level evidence from randomised clinical trials. BMJ Open. 2013 Aug 13;3(8):e003143. doi: 10.1136/bmjopen-2013-003143. PMID 23943775
- [Background] McCabe C, Claxton K, Culyer AJ. The NICE cost-effectiveness threshold: what it is and what that means. Pharmacoeconomics. 2008;26(9):733-44. doi: 10.2165/00019053-200826090-00004. PMID 18767894
- [Background] Pauker SG, Kassirer JP. Therapeutic decision making: a cost-benefit analysis. N Engl J Med. 1975 Jul 31;293(5):229-34. doi: 10.1056/NEJM197507312930505. PMID 1143303
- [Background] Hultcrantz M, Mustafa RA, Leeflang MMG, Lavergne V, Estrada-Orozco K, Ansari MT, Izcovich A, Singh J, Chong LY, Rutjes A, Steingart K, Stein A, Sekercioglu N, Arevalo-Rodriguez I, Morgan RL, Guyatt G, Bossuyt P, Langendam MW, Schunemann HJ. Defining ranges for certainty ratings of diagnostic accuracy: a GRADE concept paper. J Clin Epidemiol. 2020 Jan;117:138-148. doi: 10.1016/j.jclinepi.2019.05.002. Epub 2019 May 18. PMID 31112801
- [Background] Hultcrantz M, Rind D, Akl EA, Treweek S, Mustafa RA, Iorio A, Alper BS, Meerpohl JJ, Murad MH, Ansari MT, Katikireddi SV, Ostlund P, Tranaeus S, Christensen R, Gartlehner G, Brozek J, Izcovich A, Schunemann H, Guyatt G. The GRADE Working Group clarifies the construct of certainty of evidence. J Clin Epidemiol. 2017 Jul;87:4-13. doi: 10.1016/j.jclinepi.2017.05.006. Epub 2017 May 18. PMID 28529184
- [Background] Faraone SV. Interpreting estimates of treatment effects: implications for managed care. P T. 2008 Dec;33(12):700-11. No abstract available. PMID 19750051
- [Background] Johnston BC, Ebrahim S, Carrasco-Labra A, Furukawa TA, Patrick DL, Crawford MW, Hemmelgarn BR, Schunemann HJ, Guyatt GH, Nesrallah G. Minimally important difference estimates and methods: a protocol. BMJ Open. 2015 Oct 1;5(10):e007953. doi: 10.1136/bmjopen-2015-007953. PMID 26428330
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Guyatt GH, Thorlund K, Oxman AD, Walter SD, Patrick D, Furukawa TA, Johnston BC, Karanicolas P, Akl EA, Vist G, Kunz R, Brozek J, Kupper LL, Martin SL, Meerpohl JJ, Alonso-Coello P, Christensen R, Schunemann HJ. GRADE guidelines: 13. Preparing summary of findings tables and evidence profiles-continuous outcomes. J Clin Epidemiol. 2013 Feb;66(2):173-83. doi: 10.1016/j.jclinepi.2012.08.001. Epub 2012 Oct 30. PMID 23116689
- [Background] Baldeh T, Saz-Parkinson Z, Muti P, Santesso N, Morgano GP, Wiercioch W, Nieuwlaat R, Grawingholt A, Broeders M, Duffy S, Hofvind S, Nystrom L, Ioannidou-Mouzaka L, Warman S, McGarrigle H, Knox S, Fitzpatrick P, Rossi PG, Quinn C, Borisch B, Lebeau A, de Wolf C, Langendam M, Piggott T, Giordano L, van Landsveld-Verhoeven C, Bernier J, Rabe P, Schunemann HJ. Development and use of health outcome descriptors: a guideline development case study. Health Qual Life Outcomes. 2020 Jun 5;18(1):167. doi: 10.1186/s12955-020-01338-8. PMID 32503619
- [Background] Abramson JH. WINPEPI updated: computer programs for epidemiologists, and their teaching potential. Epidemiol Perspect Innov. 2011 Feb 2;8(1):1. doi: 10.1186/1742-5573-8-1. PMID 21288353
- [Background] Alper BS, Oettgen P, Kunnamo I, Iorio A, Ansari MT, Murad MH, Meerpohl JJ, Qaseem A, Hultcrantz M, Schunemann HJ, Guyatt G; GRADE Working Group. Defining certainty of net benefit: a GRADE concept paper. BMJ Open. 2019 Jun 4;9(6):e027445. doi: 10.1136/bmjopen-2018-027445. PMID 31167868
- [Background] Puhan MA, Singh S, Weiss CO, Varadhan R, Boyd CM. A framework for organizing and selecting quantitative approaches for benefit-harm assessment. BMC Med Res Methodol. 2012 Nov 19;12:173. doi: 10.1186/1471-2288-12-173. PMID 23163976
- [Background] Weinstein MC, Stason WB. Foundations of cost-effectiveness analysis for health and medical practices. N Engl J Med. 1977 Mar 31;296(13):716-21. doi: 10.1056/NEJM197703312961304. PMID 402576
- [Derived] Morgano GP, Mbuagbaw L, Santesso N, Xie F, Brozek JL, Siebert U, Bognanni A, Wiercioch W, Piggott T, Darzi AJ, Akl EA, Verstijnen IM, Parmelli E, Saz-Parkinson Z, Alonso-Coello P, Schunemann HJ. Defining decision thresholds for judgments on health benefits and harms using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) Evidence to Decision (EtD) frameworks: a protocol for a randomised methodological study (GRADE-THRESHOLD). BMJ Open. 2022 Mar 10;12(3):e053246. doi: 10.1136/bmjopen-2021-053246. PMID 35273045